CLINICAL TRIAL: NCT03513991
Title: Evaluation of the Impact of Infant Formulas With Different Protein Content on Growth, Gastrointestinal Tolerance, and B-casomorphin Concentration of Infants.
Brief Title: Evaluation of Different Protein Content of Formulas on Nutrition Status of Infants.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Queretaro (Other)
Collaborators: NUCITEC S.A. de C.V. (Unknown)
Responsible Party: Principal Investigator, Olga Patricia García Obregon, Principal Investigator, Universidad Autonoma de Queretaro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: F-50-02
Record Dates: First submitted 2018-04-10; First posted 2018-05-02 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Growth & Development; Formula Feeding of Healthy Full Term Infants; Breast Feeding of Healthy Full Term Infants
Keywords: human milk; infant formula with low protein; alpha lactoalbumin; growth velocity; gastrointestinal events
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Intervention Model Description: The exclusively formula-fed infants were randomized to one of three study formulas with different protein profile.
  A control group was selected with women that voluntarily chose to exclusively breast feed for at least 4 months.
Who Masked: Participant
Masking Description: The participant did not know which formula was assigned. Infant formulas were packed in the same presentation and identified by a number.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IF-VLP (very low protein) (Experimental): Participants were exclusively fed with an infant formula containing 1g of protein/dL, 26% alpha lactoalbumin, and 100% A2 casein for 4 months.
  Interventions: Other: Infant formula
- IF-LP (low protein) (Other): Participants were exclusively fed with an infant formula containing 1.3 g of protein/dL, 26% alpha lactoalbumin, 100% A2 casein for 4 months.
  Interventions: Other: Infant formula
- IF-CSP (control standard protein) (Other): Participants were exclusively fed with an infant formula containing 1.5 g of protein/dL, 50% A1 casein and 50% A2 casein for 4 months.
  Interventions: Other: Infant formula
- HM (human milk) (No Intervention): Participants were exclusively breastfed

INTERVENTIONS:
Other: Infant formula
  Arms: IF-CSP (control standard protein); IF-LP (low protein); IF-VLP (very low protein)

SUMMARY:
Human milk (HM) is the gold standard of early infant nutrition. The World Health Organization (WHO) recommend that newborns be exclusively breastfed for the first 6 months of life. It has beed reported that an exclusive breast feeding at 6 months of age range from 10 to 46%. Thus, the intake of infant formulas (IF) is quite widespread, including infants that have less than 6 months that are not receiving breast milk. Most of the commercial IF are cow's milk-based formulas that have a higher concentration of protein than breast milk and have a different protein composition. Commercial IF have a low proportion of alpha lactoalbumin, and A1 β-casein; during its digestion, a β-casomorphin 7 peptide is produced. In addition, it has a high concentration of β-lactoglobulin. Both, β-casomorphin 7 and β-lactoglobulin have been associated with a higher risk of diabetes obesity and allergies. Human β-casein does not produce β-casomorphin 7 during its digestion, it has a high concentration of alpha-lactoalbumin and does not have β-lactoglobulin.

The purpose of this study is to evaluate growth, gastrointestinal tolerance, and β-casomorphin 7 in urine of infants that are exclusively breastfed compared to infants fed three IF with different proteint content.

DETAILED DESCRIPTION:
Developing an IF with A2 β-casein, high proportion of alpha-lactoalbumin and less protein that commercial IF, similar to breast milk (1g/100 mL), could be and important strategy to decrease the risk of diseases. This infant formula was compared with breast milk and two other IF with different protein composition. The three formulas were packed in the same presentation and identified by a number. Mothers voluntarily elected to exclusively breast-feed or formula-feed her newborn. the present study

Infants' mothers were recruited from six health centers from the Health Ministry in Querétaro, México. Directors of each health center authorized the protocol study. The field workers were read and explained the informed consent letter, the objectives, procedures, risks and benefits of the study in detail.

ELIGIBILITY:
Inclusion Criteria:

* Full-term newborn (≥37 weeks of gestation)
* Birth weight ≥2500 g and ≤4000 g
* Apgar score > 8
* Infants from birth to 40 days of age at the time of enrollment
* Mothers voluntarily elected to exclusively breast-feed or formula-feed her newborn.

Exclusion Criteria:

* Infants with congenital heart defect, congenital illness or malformations, severe gastrointestinal disease, kidney, liver, central nervous system, or metabolic disease, or born from mothers with gestational diabetes.

Ages: 1 Day to 40 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2017-08-08 (Actual)

PRIMARY OUTCOMES:
Change in weight | Baseline to 4 months of age
  Weight

SECONDARY OUTCOMES:
Anthropometry measurements | Baseline, 1, 2 ,3 and 4 months of age
  Measurements will include length and head circumference, and together with the primary outcome of weight, will be used to calculate z-scores using WHO Growth Standards.
Beta-casomorphin 7 concentration | Baseline and at 4 months of age
  Quantification of beta-casomorphin 7 concentration in urine
Number of gastrointestinal events | Baseline, 1, 2, 3, and 4 months
  Gastrointestinal events will be recorded by the mothers. These events include: constipation, diarrhea, regurgitation, vomit, reflux, colic, constant crying, and stool consistency and color, using previously reported scales (Bekkali et al, 2009; Trabulsi, 2011).

CONTACTS AND LOCATIONS:
Overall Officials: Olga P Garcia, PhD, Principal Investigator — Universidad Autonoma de Queretaro
Locations (1):
- Universidad Autonoma de Queretaro, Querétaro City, Querétaro, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gonzalez-Garay AG, Serralde-Zuniga AE, Medina Vera I, Velasco Hidalgo L, Alonso Ocana MV. Higher versus lower protein intake in formula-fed term infants. Cochrane Database Syst Rev. 2023 Nov 6;11(11):CD013758. doi: 10.1002/14651858.CD013758.pub2. PMID 37929831